CLINICAL TRIAL: NCT04129203
Title: Multi Center, Prospective, Registry Trial of Versi Retriever Mechanical Thrombecomy for Acute Ischemic Stroke in Japan
Brief Title: Versi Retriever Approving Trial in Japan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kobe City General Hospital (Other)
Responsible Party: Principal Investigator, Nobuyuki Sakai, Director, Neurosurgery, Kobe City General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-01
Record Dates: First submitted 2019-03-12; First posted 2019-10-16 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Stroke, Acute
Keywords: acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial arm (Experimental): Mechanical thrombectomy using Versi Retriever
  Interventions: Device: Versi Retriever thrombectomy

INTERVENTIONS:
Device: Versi Retriever thrombectomy — Mechanical thrombectomy using Versi Retriever

SUMMARY:
This is Versi Retriever mechanical thrombectomy device approving study in Japan. Multi center, single arm, prospective registry trial. Physicians control trial, conducted my N Sakai, Kobe City Medical Center General Hospital.

DETAILED DESCRIPTION:
This is Versi Retriever mechanical thrombectomy device approving study in Japan. Multi center, single arm, prospective registry trial. Physicians control trial, conducted my N Sakai, Kobe City Medical Center General Hospital.

60 cases will be enrolled and 90 days follow up need. Primary endpoint is favorable clinical outcome, mRS 0-2. Secondary endpoint are mortality in 90days, immediate successful recanalization, TICI 2b-3, symptomatic intracranial hemorrhage, and any adverse event related to device and or procedure.

ELIGIBILITY:
Inclusion Criteria:

* acute onset neurological sympto m related to occluded vessel
* within 8 hours from onset to tre atment or within 24 hours from onset to treatment with imaging diagnosis
* contra-indication or failed to int ravenous rt-PA
* accessible occlusion at ICA, MC A, VA, BA, PCA
* 5-30 of NIHSS
* 0-2 of mRS before onset
* obtain documented informed co ntent

Exclusion Criteria:

* following condition; arterial diss ection, engird, inaccessible turtuousity, difficult access by 50% or m ore stenosis, acute intracranial hemorrhage, space occuping lesion or brain tumor, major early ischemic change in brain
* occlude 2 major vessel territory
* allege for contrast media,
* abnormal PTT/APTT within 4 h ours intravenous heparin
* hemorrhagic tendency or 3 or more INR with Warfarin administration
* 30000cc or less of Platelet
* 50mg/dL or less of blood sugar
* uncontrolled blood pressure, 185mmHg or more at systolic, 110m mHg or more at diastolic
* 90days or less life expancy
* pregnant or lactating
* join another trial of medicine or medical device
* ineligible for trial

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Good clinical outcome | 90days after procedure
  modified Rankin Score is 0-2

SECONDARY OUTCOMES:
Successful recanalization | at 3 passes of device in the procedure
  TICI 2b-3
Successful recanalization | at end of procedure
  TICI 2b-3
Symptomatic and asymptomatic intracranial hemorrhage | at 24 hours after procedure
  NIHSS 4 or more worsened
Good clinical outcome 2 | 90days after procedure
  mRS 0-2 or NIHSS 10 or more improvement
sever advers event | 90days after procedure
  device or procedure related

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sakai, MD DMSc, Study Chair — Kobe City Medical Center General Hospital
Locations (1):
- Kobe City Medical Center General Hospital, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No